CLINICAL TRIAL: NCT05434702
Title: The "COACH" Study: Individualized COaching in Young Adult Cancer Survivors to Encourage Healthy Behaviors
Brief Title: "COACH" Study: Individualized COaching in Young Adult Cancer Survivors to Encourage Healthy Behaviors
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-21786; R03CA270475 (NIH)
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Health Behavior
Keywords: Young Adult; Cancer survivor
MeSH Terms: conditions — Health Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adult cancer survivors: Adolescent and young adult cancer survivors
  Interventions: Behavioral: Digital Diet Diary; Behavioral: NHANES Food Frequency Questionnaire (FFQ); Behavioral: Fitbit data collection; Behavioral: Quality of Life questionnaire; Behavioral: Functional Assessment of Cancer Therapy - General (FACT-G) Questionnaire; Behavioral: Godin Exercise Leisure-Time questionnaire; Behavioral: Zoom interviews

INTERVENTIONS:
Behavioral: Digital Diet Diary — Participants will be asked to complete the Fitbit 3-day food record, which consists of inputting each food and beverage consumed for two weekdays and 1 weekend day into the Fitbit application. This digital diary includes taking photos of each food and beverage consumed during the 3 day food record period on the participant's iphone or ipad.
Behavioral: NHANES Food Frequency Questionnaire (FFQ) — Participants will complete the the Food Frequency questionnaire which indicates usual food intake over the past year.
Behavioral: Fitbit data collection — Participants will be asked to wear a Fitbit continuously (24/7) for one week to track steps and activity intensity. The Fitbit is worn on the wrist and uses accelerometer and heart rate technology to quantify steps taken and integrated barometric altimeter to measure activity intensity. The resulting Fitbit data will be automatically pulled from the participant's smartphone or study device.
Behavioral: Quality of Life questionnaire — The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) includes questions about participant's quality of life during the past week, self-reported general health, self reported chronic conditions and psychological distress using a scale from 1-5, 1=excellent, 5= poor. A lower total score indicates better qualify of life.
Behavioral: Functional Assessment of Cancer Therapy - General (FACT-G) Questionnaire — The Functional Assessment of Cancer Therapy - General (FACT-G) Questionnaire includes questions about participant's physical, social, emotional and functional well being over the past 7 days. This questionnaire uses a 5 point Likert-type scale, 0=not at all, 4=very much. A higher total score indicates better quality of life.
Behavioral: Godin Exercise Leisure-Time questionnaire — The Godin Exercise Leisure-Time questionnaire measures the frequency of strenuous, moderate, and mild exercise for periods of 15 minutes or more during the participant's free time throughout a typical week. The scoring using the formula leisure score index (LSI) which is obtained using the following formula: (frequency of mild × 3) + (frequency of moderate × 5) + (frequency of strenuous × 9).
Behavioral: Zoom interviews — A subset of 30 participants (10 African American, 10 Hispanic, 10 non-Hispanic white) will participate in semi-structured interviews to explore (a) sociocultural, environmental, and individual factors associated with lifestyle behaviors; (b) awareness of American Cancer Society (ACS) guidelines, current practices, and essential intervention modules (ex. integrating cultural foods and preferences) to provide study team with information needed to develop healthy behavior interventions for young adult cancer survivors.

SUMMARY:
The purpose of this study is to better understand the current lifestyle behaviors that people with a young adult cancer diagnosis have after treatment. Investigators are also interested in understanding what affects the quality of life of young adult cancer survivors. Investigators will use this information to develop and test a diet and physical activity intervention to help young adult cancer survivors feel their best

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer between the ages of 19 and 29
* Currently between the ages of 20 and 30 years old
* At least 1 year post-adjuvant therapy
* Able to read/speak English
* Able to complete an online survey
* Able to consume food orally

Exclusion Criteria:

* Women who are pregnant

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primarily participants in Moffitt Cancer Center's Adolescent and Young Adult Survivorship program
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Quality of Life in YA Cancer Survivors -EORTC-QOL | Week 1
  Quality of life will be measured using the EORTC-QOL questionnaire. The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) includes questions about participant's quality of life during the past week, self-reported general health, self reported chronic conditions and psychological distress using a scale from 1-5, 1=excellent, 5= poor. A lower total score indicates better qualify of life
Aim 1: Quality of Life in YA Cancer Survivors -FACT-G | Week 1
  Quality of life will be measured using the FACT-G questionnaire. The Functional Assessment of Cancer Therapy - General (FACT-G) Questionnaire includes questions about participant's physical, social, emotional and functional well being over the past 7 days. This questionnaire uses a 5 point Likert-type scale, 0=not at all, 4=very much. A higher total score indicates better quality of life.
Aim 1: Physical Activity in YA cancer Survivors - Questionnaire | Up to 2 weeks
  Frequency and intensity of physical activity will be measured using the Godin Exercise leisure time questionnaire. The Godin Exercise Leisure-Time questionnaire measures the frequency of strenuous, moderate, and mild exercise for periods of 15 minutes or more during the participant's free time throughout a typical week. The scoring using the formula leisure score index (LSI) which is obtained using the following formula: (frequency of mild × 3) + (frequency of moderate × 5) + (frequency of strenuous × 9).
Aim 1: Physical Activity in YA cancer Survivors - Fitbit data | Up to 2 weeks
  Frequency and intensity of physical activity will be measured using Fitbit data.
Aim 1: Healthy eating in YA cancer survivors | Up to 2 weeks
  Data from the the food frequency questionnaire along with digital diet diary will be compared to American Cancer Society dietary guidelines.

SECONDARY OUTCOMES:
Aim 2: Development of educational intervention for YA cancer survivors | Up to 24 months
  Data collected from zoom interviews with a sub-set participants will be used to provide study team with information needed to develop healthy behavior interventions for young adult cancer survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Heather S.L. Jim, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE